CLINICAL TRIAL: NCT03963908
Title: Evidence-based Pain Intervention for Veterans: Leveraging Mobile & Social Media: A Randomized 262-subject Controlled Trial of AtEase, a Pain Self-management App in the Treatment of Chronic Pain in Veterans
Brief Title: Evidence-based Pain Intervention for Veterans: AtEase for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Principal Investigator, Sara Johnson, Co-President & CEO, Pro-Change Behavior Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9R44AT009675-02 (NIH)
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Chronic Pain
Keywords: chronic pain; stage of change; pain self management; mobile applications; Transtheoretical Model
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This study involves a 2-group X 3 occasion randomized trial that will examine whether AtEase produces more significant improvements in PEG scores (which reflect total pain intensity and pain interference) than a comparison intervention (i.e., an existing online pain self-management intervention entitled Chronic Pain Education for Veterans).
Who Masked: Participant
Masking Description: Participants will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): AtEase is a mobile app designed to promote pain self-management, healthy sleep habits, and effective stress management. It includes a tailored Newsfeed that updates regularly with articles, activities, videos, and quizzes chosen for the user; a chat feature that asks questions and provide tailored feedback; a Message Center; and a Pain Tracker. Users can interact with AtEase as often as they like for six months.
  Interventions: Behavioral: AtEase
- Comparison (Active Comparator): Chronic Pain Education for Veterans is a VA-endorsed pain management online educational curriculum that provides CBT pain self-management materials. Users randomized to the comparison condition will have unlimited access for 6 months.
  Interventions: Behavioral: Chronic Pain Education

INTERVENTIONS:
Behavioral: AtEase — AtEase is a tailored pain self-management mobile app that tailors participant's feedback based on readiness to engage in pain self-management and preference for self-management strategies.
  Arms: Intervention
Behavioral: Chronic Pain Education — CBT-based Education on Pain Self-Management for Veterans
  Arms: Comparison

SUMMARY:
This study is a randomized controlled trial to test the efficacy AtEase, a pain self-management app in a sample of Veterans with chronic musculoskeletal pain. The primary outcome is changes in PEG scores from baseline to final follow-up (12 months).

DETAILED DESCRIPTION:
The primary objectives of this project are to develop and examine the effectiveness of a mobile app (AtEase) that is designed to provide tailored behavior change guidance to promote pain self-management, healthy sleep habits, and effective stress management in a randomized clinical trial including 262 Veterans with chronic pain.

Veterans will be recruited from VA Connecticut Healthcare, as well as from numerous diverse community recruitment channels (including employers, community groups that provide services for Veterans, Student Veterans of America, and social media).

Eligible Veterans will be randomized to receive access to AtEase or the comparison intervention (a mobile-optimized adaptation of Chronic Pain Education for Veterans) for a total of 6 months. AtEase is a tailored pain self-management mobile app that tailors participant's feedback based on readiness to engage in pain self-management and preference for self-management strategies. Chronic Pain Education for Veterans is a free VA-endorsed publicly available pain management online educational curriculum that provides cognitive-behavioral therapy-based pain self-management materials.

Between the baseline assessment and the 6-month follow up assessment, participants will have unlimited access AtEase or the Chronic Pain Education for Veterans program. All participants will complete follow-up assessments at 6 months and 12-months post-baseline.

The primary outcome will be a comparison of PEG scores at 12 months follow-up. Secondary outcomes will include pain,Global Impression of Change; readiness to self-manage pain, manage stress, and engage in healthy sleep habits; well-being; and Post Traumatic Stress Disorder Checklist scores.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Veteran
* Chronic musculoskeletal pain defined as (numeric rating scale of >4) (10 point scale) for > 3 months.43
* Internet connectivity via tablet or mobile phone.

Exclusion Criteria:

* Life-threatening condition or acute medical conditions that precludes participation
* Psychiatric conditions that could impair participation
* Suicidal ideation or intent
* Inability to read or speak English
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
PEG | Baseline to 12 months
  The PEG is a multi-dimensional three-item assessment that measures average pain rating, as well as both emotional and physical functioning.

SECONDARY OUTCOMES:
Global Impression of Change | 12 months
  The Global Impression of Change scale is recommended43 as a core outcome measure in pain studies. It is a single item that asks participants to describe any change in their condition as a result of using the program. Response options range from 1 = No change (or condition has gotten worse) to 7 = A great deal better, and a considerable improvement that has made all the difference.
Pain Level | Baseline to 12 months
  Level of pain will also be assessed by asking participants to rate their pain 1) right now, 2) usual level of pain in the last week, 3) best level of pain in the last week, and 4) worst level of pain in the last week. All ratings are on a scale of 0-10, with zero equal to no pain, and 10 equal to worst pain.
Readiness to self-manage pain | Baseline to 12 months
  Changes in participant's stage of change for using self-management strategies using a stage of change algorithm
Stage of change for healthy sleep habits | Baseline to 12 months
  Readiness to get at least 7 hours of sleep a night
Stage of change for stress management | Baseline to 12 months
  Readiness to effectively manage stress
Post-Traumatic Stress Disorder (PTSD) Checklist (PCL-5) | Baseline to 12 months
  PTSD symptoms will be measured using the 20-item PCL-5, which assesses the 20 symptoms of PTSD.
Well-Being | Baseline to 12 months
  Well-being will be assessed using the Cantril Self-Anchoring Scale, which asks participants to imagine a ladder with steps numbered from 0 to 10, with the top representing the best possible life and the bottom representing the worst possible life. Participants indicate where they feel their life falls currently and where it will fall in five years.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Johnson, PhD, Principal Investigator — Pro-Change Behavior Systems, Inc.
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Pro-Change Behavior Systems, Inc, South Kingstown, Rhode Island

IPD SHARING:
Plan to Share IPD: No